CLINICAL TRIAL: NCT00089440
Title: Assessment of Interactions Between IV Methamphetamine and Aripiprazole
Brief Title: Assessment of Interactions Between Methamphetamine and Aripiprazole - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-MDS-0002-1
Record Dates: First submitted 2004-08-05; First posted 2004-08-06 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-07

CONDITIONS: Amphetamine-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The purpose of this study is to assess the interactions between intravenous methamphetamine and aripiprazole.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled human laboratory clinical pharmacology study to assess potential interactions between intravenous d-methamphetamine infusion and treatment with oral aripiprazole.

ELIGIBILITY:
Inclusion Criteria:

* Must meet DSM-4 criteria for methamphetamine abuse or dependence and are non-treatment seeking.
* Ability to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.

Exclusion Criteria:

* Please contact the site for more information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17
Dates: Start 2004-06; Study Completion 2005-03

PRIMARY OUTCOMES:
Adverse effect measures
pharmacokinetic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Newton, M.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA Integrated Substance Abuse Program, Los Angeles, California
  - New York University, School of Medicine, New York, New York